CLINICAL TRIAL: NCT04412304
Title: Patient Characteristics, Outcome and Thromboembolic Events Among Adult Critically Ill COVID-19 Patients With Different Anticoagulant Regimes at One of the Biggest Emergency Hospitals in Northern Europe, Sweden
Brief Title: Anticoagulant Therapy and 28-days Mortality in Critically Ill COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Christer Svensen, Professor, Karolinska Institutet
Other Study IDs: Anticoagulant therapy Covid-19
Record Dates: First submitted 2020-05-30; First posted 2020-06-02 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Covid-19; Thromboembolic Events; Bleeding
MeSH Terms: conditions — COVID-19; Thromboembolism; Hemorrhage | interventions — Dalteparin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- thrombose prophylaxis: The dose used to prevent thromboembolic complication in critically ill
  Interventions: Drug: Dose of Tinzaparin or Dalteparin
- double thrombose prophylaxis: Double the dose used to prevent thromboembolic complication in critically ill
  Interventions: Drug: Dose of Tinzaparin or Dalteparin
- full dose anticoagulant: Dose used to treat thromboembolic event
  Interventions: Drug: Dose of Tinzaparin or Dalteparin

INTERVENTIONS:
Drug: Dose of Tinzaparin or Dalteparin — The patients will be categorised into three groups depending on initial regime of anticoagulants after arrival in the ICU.

SUMMARY:
The aims of the study are to to associate anticoagulation (AC) regime with outcome in critically ill patients with Covid-19. This will be done by describe baseline characteristics and comorbidities before hospital admission, level of organ support and dose of AC treatment and associate this with 28 days survival, survival outside ICU, thromboembolic event and bleeding complications.

ELIGIBILITY:
Inclusion Criteria:

* laboratory confirmed positive test for SARS-CoV-2
* admitted to ICU because of critical illness due to covid-19

Exclusion Criteria:

* patients with treatment for thromboembolic complications at arrival to the ICU
* short ICU length of stay defined as discharged the same or the following day as ICU admission

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A cohort study of the Covid-19 patients admitted to an ICU at Stockholm South General Hospital from March 6th 2020 to April 30 2020
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
28-days ICU mortality | 28 days from ICU-admission
  28-days ICU mortality from admission to the ICU. Discontinue of ICU-care to palliative care counts as death.

SECONDARY OUTCOMES:
Incidence of thromboembolic events | 28 days from ICU-admission
  Thromboembolic events are defined as pulmonary emboli (PE), deep venous thrombus (DVT), ischemic stroke and other peripheral arterial emboli. PE is defined as PE verified by computer tomography or by findings of acute strain of the right heart on echocardiography combined with a clinical interpretation of the patients deteriorating as a probable PE stated in the medical records. DVT is defined as DVT verified with ultrasound. Ischemic stroke is defined as ischemic stroke verified by computer tomography. Peripheral arterial emboli are defined as peripheral arterial emboli verified by computer tomography.
Incidence of bleeding events | 28 days from ICU-admission
  The event of bleeding will be defined by WHO modified bleeding scale as 1-4.
ICU-free days alive from ICU-admission. | 28 days from ICU-admission
  ICU-free days alive during 28 days from ICU-admission. Counts as 0 days if discharged to ward for palliative treatment.

OTHER OUTCOMES:
D-dimer levels in the three groups groups | 28 days from ICU-admission
  D-dimer every day it is measured during first 28 days from ICU-admission.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cronhjort, PhD, Principal Investigator — Karolinska Institutet, Department of Clinical Science and Education
Locations (1):
- South General Hospital, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Derived] Jonmarker S, Hollenberg J, Dahlberg M, Stackelberg O, Litorell J, Everhov AH, Jarnbert-Pettersson H, Soderberg M, Grip J, Schandl A, Gunther M, Cronhjort M. Dosing of thromboprophylaxis and mortality in critically ill COVID-19 patients. Crit Care. 2020 Nov 23;24(1):653. doi: 10.1186/s13054-020-03375-7. PMID 33225952